CLINICAL TRIAL: NCT06423326
Title: A Single-Arm Phase II Clinical Trial of Gemcitabine, Cisplatin, and Nab-Paclitaxel as Neoadjuvant Therapy for Pancreatic Ductal Adenocarcinoma
Brief Title: Gemcitabine, Cisplatin and Nab-Paclitaxel as Neoadjuvant Treatment for Patients With Resectable or Borderline Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mihir M. Shah, MD, FACS, FSSO, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006976; NCI-2024-02082 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP6093-23 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); STUDY00006976 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2024-04-10; First posted 2024-05-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Borderline Resectable Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Adenocarcinoma; Stage I Pancreatic Cancer AJCC v8; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Magnetic Resonance Spectroscopy; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nab-paclitaxel, cisplatin, gemcitabine) (Experimental): Patients receive nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 15 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease, partial or complete response undergo surgical resection per standard of care. Additionally, patients undergo biopsy on study and undergo blood sample collection and CT or MRI at pre-study and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Drug: Nab-paclitaxel; Procedure: Pancreatic Surgical Procedure

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
Procedure: Pancreatic Surgical Procedure — Undergo surgical resection
  Other Names: Pancreatic Surgery

SUMMARY:
This phase II trial tests how well gemcitabine, cisplatin and nab-paclitaxel given before surgery (neoadjuvant) works in treating patients with pancreatic cancer that can be removed by surgery (resectable) or that is borderline resectable. The standard treatment for resectable and borderline resectable pancreatic cancer is a combination of surgery and chemotherapy. Neoadjuvant therapy has been shown to improve overall survival compared to patients receiving surgery first. Gemcitabine is a chemotherapy drug that blocks the cells from making DNA and may kill tumor cells. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Nab-paclitaxel is an albumin-stabilized nanoparticle formulation of paclitaxel, an antimicrotubule agent that stops tumor cells from growing and dividing and may kill them. Nab-paclitaxel may have fewer side effects and work better than other forms of paclitaxel. Gemcitabine, cisplatin and nab-paclitaxel may be an effective neoadjuvant treatment option for patients with resectable or borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the major pathological response rate, feasibility and safety of biweekly gemcitabine, cisplatin and nab-paclitaxel (GCN) in the neoadjuvant setting for patients with resectable and borderline resectable pancreatic ductal adenocarcinoma.

SECONDARY OBJECTIVE:

I. Determine if neoadjuvant GCN increases tumoral infiltration of lymphocytes with local and systemic phenotypic features that assist in the antitumor immune response.

OUTLINE:

Patients receive nab-paclitaxel intravenously (IV) over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 15 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease, partial or complete response undergo surgical resection per standard of care. Additionally, patients undergo biopsy on study and undergo blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) at pre-study and on study.

After completion of study treatment, patients are followed up every 3-4 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed - resectable and borderline resectable pancreatic ductal adenocarcinoma

  * Resectability will be defined as per National Comprehensive Cancer Network (NCCN) guidelines using cross-sectional imaging (contrast-enhanced computed tomography or magnetic resonance imaging scans of the abdomen, and pelvis)
  * Decisions about resectability status will be made in consensus at multidisciplinary meetings/discussions

Resectable disease will be defined as:

* No interface of the tumor with celiac artery, common hepatic artery (CHA), or superior mesenteric arteries (SMA) (and, if present, variants)
* Less than 180° interface between tumor and vessel wall of the portal or superior mesenteric veins (SMV) without vein contour irregularity
* For tumors of the body and tail of the pancreas, interface with the splenic artery and splenic vein of any degree will be considered resectable disease

Borderline resectable disease will be defined as:

* To include at least one of the following:

  * Tumor abutment < 180° of the superior mesenteric artery or celiac axis
  * Solid tumor contact with CHA without extension to celiac artery (CA) or hepatic artery bifurcation allowing for safe and complete resection and reconstruction
  * Solid tumor contact with variant arterial anatomy (ex: accessory right hepatic artery, replaced right hepatic artery, replaced CHA, and the origin of replaced or accessory artery)
  * Tumor induced narrowing of SMV, portal vein (PV) or SMV-PV of > 180˚ of the diameter of the vessel
  * Short segment occlusion of the SMV, PV or SMV-PV with a suitable PV above and SMV below, for reconstruction
  * Solid tumor contact with inferior vena cava
  * Biopsy proven N1 disease (regional lymph nodes involved) from pre-referral biopsy or endoscopic ultrasound (EUS)-guided fine needle aspiration (FNA)

    * No distant extrapancreatic disease (M0)
    * Adults > 18 years of age
    * Able to give informed consent
    * Able to adhere to study visit schedule and other protocol requirements
    * Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
    * Absolute neutrophil count (ANC) ≥ 1,500 cells/ul
    * Platelet count ≥ 100,000 cells/ul
    * Hemoglobin ≥ 9 g/dL
    * Serum total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
    * Albumin ≥ 3 g/dl
    * Creatinine ≤ 1.5 x ULN
    * Male, or a non-pregnant and non-lactating female
    * Women of child-bearing potential - defined as a sexually mature woman who has not undergone hysterectomy - the surgical removal of the uterus or bilateral oophorectomy - the surgical removal of both ovaries or has not been naturally postmenopausal for at least 24 consecutive months, i.e., has had menses at any time during the preceding 24 consecutive months, must commit to true abstinence from heterosexual contact, or agree to use, and be able to comply with, effective contraception without interruption for 28 days prior to starting gemcitabine/cisplatin/nab- paclitaxel (including dose interruptions) until treatment with gemcitabine/cisplatin/nab-paclitaxel is complete
    * Male subjects must practice true abstinence or agree to use a condom during sexual contact with a female of childbearing potential or a pregnant female while on treatment (including during dose interruptions) with gemcitabine/cisplatin/nab-paclitaxel and for 6 months following gemcitabine/cisplatin/nab- paclitaxel discontinuation, even if he has undergone a successful vasectomy

Exclusion Criteria:

* Peripheral neuropathy of grade 2 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 4.0. In CTCAE version 4.0 grade 2 sensory neuropathy is defined as "moderate symptoms; limiting instrumental activities of daily living (ADLs)"
* Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, symptomatic congestive heart failure, uncontrolled diabetes, serious active, uncontrolled infection after inadequate biliary drainage if tumor obstructing bile duct, or psychiatric illness/social situations
* Pregnancy (positive pregnancy test) or lactation
* Known central nervous system (CNS) disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (radiosurgery [RS]; Gamma Knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded
* Previous (within the past 5 years) or concurrent presence of other untreated cancer, except nonmelanoma skin cancer and in situ carcinomas
* History of allergy or hypersensitivity to any of the study drugs
* Current abuse of alcohol or illicit drugs
* Inability or unwillingness to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Response Rate to Neoadjuvant Chemotherapy | Up to 24 months
  Clinical response is defined as biochemical, radiological, pathological response or stable disease. • Biochemical response (or CA 19-9 response) is defined as >50% decrease from baseline with tumor response. Radiologic response is defined as complete response (CR), partial response (PR) or stable disease (SD) after the neoadjuvant therapy per RECIST 1.1. Pathologic response is defined by CAP scoring system as 0 (complete response), 1 (moderate response), 2 (minimal response) and 3 (poor or no response). Stable disease is defined as the absence of biochemical response (>50% CA 19-9 reduction), radiological response (per RECIST 1.1), or major pathological response (CAP Score 0-1), without metastasis / unresectability, and patient undergoes surgical resection. Clinical response rate (including clinical, biochemical, radiological, pathological response or stable disease) will be reported as a proportion, with an exact 90% confidence interval estimated using the Clopper-Pearson method.

SECONDARY OUTCOMES:
Treatment Completion | Up to 24 months
  Feasibility will be defined as completion of all preoperative and operative therapy. Treatment completion will reported as a proportion, with an exact 95% confidence interval estimated using the Clopper-Pearson method.
Incidence of Adverse Events (AEs) | Up to 28 days after last dose of study treatment
  AEs, with severity will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Descriptive statistics will be reported, using frequencies and percentages for each toxicity.
Radiologic Response Rate | Up to 24 months
  Radiological response rate will be defined as complete response, partial response or stable disease after study treatment evaluated using Response Evaluation Criteria in Solid Tumors version 1.1. Radiologic response rate will be reported as a proportion, with an exact 95% confidence interval estimated using the Clopper-Pearson method.
Pathological Response Rate | Up to 24 months
  To assess the major pathological response rate (CAP 0-1) in the surgical resection specimen
Neoadjuvant Systemic Chemotherapy Rate | Up to 4 months
  To assess the rate of neoadjuvant systemic chemotherapy completion (Duration 4 months) without dose reduction
R0 Resection Rate | At time of surgery
  R0 resection indicates a microscopically margin-negative resection. R0 resection rate will reported as a proportion, with an exact 95% confidence interval estimated using the Clopper-Pearson method.
Nodal Status | Up to 24 months
  N0, N1, and N2 will be reported using frequencies and percentages.
Recurrence-Free Survival (RFS) | From surgery to recurrence or death, assessed up to 24 months
  RFS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median RFS will be estimated using the Brookmeyer-Crowley approach.
Overall Survival (OS) Rate | From study treatment start to date of death, assessed up to 24 months
  OS will be estimated using the Kaplan-Meier method, and median survival will be calculated. A 95% confidence interval will be estimated using the Brookmeyer-Crowley approach.
Carbohydrate Antigen (CA)19-9 response | Up to 24 months
  CA19-9 response will be defined as > 50% decrease from baseline will be correlated with tumor response. CA19-9 will be reported as a proportion, with an exact 95% confidence interval estimated using the Clopper-Pearson method. CA19-9 will be correlated with RFS and OS using log-rank tests and Cox proportional hazards regression. Model assumptions will be checked and verified.

CONTACTS AND LOCATIONS:
Overall Officials: Mihir M Shah, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States